CLINICAL TRIAL: NCT03124875
Title: Pilot Study to Investigate Safety, Effectiveness and Feasibility of LimFlow Stent Graft System for Creating an AV Fistula for the Treatment of Critical Limb Ischemia
Brief Title: PROMISE I Early Feasibility Trial of the LimFlow Stent Graft System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LimFlow, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECO-02527-009
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Critical Limb Ischemia; Chronic Limb-Threatening Ischemia
Keywords: Transcatheter Arterialization of Deep Veins; Percutaneous Deep Vein Arterialization; LimFlow System
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): Treated with the LimFlow System
  Interventions: Device: LimFlow System

INTERVENTIONS:
Device: LimFlow System — Creation of an AV fistula in below-the-knee vasculature for the treatment of critical limb ischemia.

SUMMARY:
This pilot study will investigate the safety, effectiveness and feasibility of the LimFlow Stent Graft System for creating an AV fistula in the Below The Knee (BTK) vascular system using an endovascular, minimally invasive approach for the treatment of Critical Limb Ischemia (CLI) in subjects ineligible for conventional endovascular or surgical limb salvage procedures.

DETAILED DESCRIPTION:
The PROMISE I Trial was a prospective, multi-center, single-arm, investigational feasibility study assessing the LimFlow System for the treatment of chronic- limb-threatening ischemia by creating an arterio-venous fistula in the below-the-knee vasculature. The study was run under an investigational device exemption (IDE G160156, NCT03124875).

Thirty-two subjects were enrolled under protocol revisions A, B, C, and D at seven sites in the United States between 5-July-2017 and 8-April-2019.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of critical limb ischemia with hemodynamic evidence of severely diminished arterial inflow of the index limb and Rutherford Classification 5 r 6
* Reviewed and approved for eligibility by the Investigator and the Independent Safety Committee (ISC)

Exclusion Criteria:

* Concomitant hepatic or renal insufficiency, thrombophlebitis, deep venous thrombus, coagulation disorder
* Severe heart failure, recent MI or stroke
* Significant peripheral edema or infection that may preclude insertion of a prosthesis or significantly impair wound healing
* Known allergies or contraindications to anti platelet therapy or device materials
* Immunodeficiency disorder or immunosuppressant therapy
* Life expectancy < 12 months

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2021-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jihad Mustapha, MD, Principal Investigator — Metro Health, University of Michigan
Locations (7):
- United States (7):
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Kaiser Permanente, Honolulu, Hawaii
  - Metro Health, University of Michigan, Wyoming, Michigan
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Mount Sinai Health System, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Palmetto Health, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mustapha JA, Saab FA, Clair D, Schneider P. Interim Results of the PROMISE I Trial to Investigate the LimFlow System of Percutaneous Deep Vein Arterialization for the Treatment of Critical Limb Ischemia. J Invasive Cardiol. 2019 Mar;31(3):57-63. doi: 10.25270/jic/18.00340. PMID 30819976
- [Result] Clair DG, Mustapha JA, Shishehbor MH, Schneider PA, Henao S, Bernardo NN, Deaton DH. PROMISE I: Early feasibility study of the LimFlow System for percutaneous deep vein arterialization in no-option chronic limb-threatening ischemia: 12-month results. J Vasc Surg. 2021 Nov;74(5):1626-1635. doi: 10.1016/j.jvs.2021.04.057. Epub 2021 May 18. PMID 34019990

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (13.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 19
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 32
Baseline Rutherford Class 5 [Count of Participants; unit: Participants] — Minor tissue loss - non-healing ulcer, focal gangrene with diffuse pedal ischemia.
  Participants | 28
Baseline Rutherford Class 6 [Count of Participants; unit: Participants] — Major tissue loss - extending above transmetatarsal level, functional foot no longer salvageable
  Participants | 4

OUTCOME MEASURES:

1. Primary Outcome: Amputation-free Survival
Description: Percentage of subjects with freedom from above-ankle amputation of the index limb and freedom from all-cause mortality
Time Frame: 30 days post-procedure
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 32
Percentage of participants | 90.6 [73.7 to 96.9]

2. Secondary Outcome: Amputation-free Survival
Description: Percentage of subjects with freedom from above-ankle amputation of the index limb and freedom from all-cause mortality
Time Frame: 6 months post-procedure
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 32
Percentage of participants | 73.8 [54.4 to 86.0]

3. Secondary Outcome: Primary Patency
Description: Percentage of patients with absence of total occlusion of the stent graft without prior clinically-driven major re-intervention of the stent graft. Total occlusion is defined as absence of flow on color doppler or angiogram and clinically-driven major re-intervention is defined as creation of a new surgical bypass, use of thrombectomy or thrombolysis, or major surgical revision performed for occlusion of the stent graft.
Time Frame: 30 days post-procedure
Population: Population analyzed was those patients that successfully underwent the index procedure. One patient did not have procedural success resulting in n=31
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 31
Percentage of participants | 73.2

4. Secondary Outcome: Primary Patency
Description: Percentage of patients with absence of total occlusion of the stent graft without prior clinically-driven major re-intervention of the stent graft.Total occlusion is defined as absence of flow on color doppler or angiogram and clinically-driven major re-intervention is defined as creation of a new surgical bypass, use of thrombectomy or thrombolysis, or major surgical revision performed for occlusion of the stent graft.
Time Frame: 6 months post-procedure
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 31
Percentage of participants | 29.3

5. Secondary Outcome: Secondary Patency
Description: Percentage of patients with absence of total occlusion of the stent graft with or without prior clinically-driven major re-intervention of the stent graft.Total occlusion is defined as absence of flow on color doppler or angiogram and clinically-driven major re-intervention is defined as creation of a new surgical bypass, use of thrombectomy or thrombolysis, or major surgical revision performed for occlusion of the stent graft.
Time Frame: 6 months post-procedure
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 31
Percentage of participants | 49.5

6. Secondary Outcome: Limb Salvage
Description: Percentage of subjects with freedom from above-ankle amputation of the index limb
Time Frame: 12 months post-procedure
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 31
Percentage of participants | 75.9 [55.8 to 87]

7. Secondary Outcome: Wound Healing
Description: Percentage of subjects with full wound healing
Time Frame: 12 months post-procedure
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 31
Percentage of participants | 58.7

8. Secondary Outcome: Deterioration in Renal Function
Description: Percentage of subjects with a 25% increase in serum creatinine after using iodine contrast agents, without another clear cause for kidney injury.
Time Frame: 6 months post-procedure
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 31
Percentage of participants | 9.4

9. Secondary Outcome: Technical Success
Description: Percentage of subjects with completion of the endovascular procedure and immediate morphological success with successful placement of the arterial and venous catheters in the desired location in the limb, and ability to place the stent graft.
Time Frame: Post-procedure, immediately
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 32
Percentage of participants | 96.9

10. Secondary Outcome: Procedural Success
Description: Percentage of subjects with a combination of Technical Success and absence of all-cause mortality, above-ankle amputation or clinically driven major re-intervention of the stent graft.
Time Frame: 30 days post-procedure
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 32
Percentage of participants | 77.4

ADVERSE EVENTS:
Time Frame: All-Cause Mortality (as a component of amputation-free survival) assessed up to 6 months. Serious and Other Adverse Events assessed to 30 days.
Description: All adverse events were reviewed by an independent Medical Monitor to determine whether an event met the trigger for adjudication by Independent Clinical Events Committee for the following endpoints: all-cause mortality, amputation documented at ankle or above, target limb thrombosis or occlusion, target limb reintervention, or deterioration in renal function.
Groups:
- Treatment: Treated with the LimFlow Stent Graft System
  LimFlow Stent Graft System: Creation of an AV fistula in below-the-knee vasculature for the treatment of critical limb ischemia.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 19/32
Other Adverse Events (participants affected / at risk) | 16/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=32)
Access Site Bleeding Requiring Transfusion (Injury, poisoning and procedural complications) | 2 (2)
Edema (Vascular disorders) | 1 (1)
Ischemia, Target Limb (Failed Procedure) (Vascular disorders) | 1 (1)
Non-Study Device Balloon Rupture and Embolization Requiring Additional Treatment/Stenting (Injury, poisoning and procedural complications) | 1 (1)
Vessel Occlusion/Thrombus Formation (Vascular disorders) | 7 (7)
Wound Bleeding or Requiring Debridement (Skin and subcutaneous tissue disorders) | 1 (1)
Wound Infection, New or Worsening (Infections and infestations) | 6 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=32)
Access Site Pain or Oozing (Injury, poisoning and procedural complications) | 2 (2)
Acute Heart Failure (Cardiac disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Arrhythmia (Cardiac disorders) | 2 (2)
Deterioration in Renal Function (Renal and urinary disorders) | 1 (1)
Edema (Vascular disorders) | 2 (2)
HyperGlyemia (Endocrine disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Immediate Post Procedure Edema (Vascular disorders) | 2 (2)
Mental Status Changes (Psychiatric disorders) | 2 (2)
New Wound on Target Limb (Skin and subcutaneous tissue disorders) | 1 (1)
Pain, Target Limg (Vascular disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Post-Procedure Anemia (Blood and lymphatic system disorders) | 1 (1)
Rectal Prolapse (Gastrointestinal disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Vessel Occlusion/Thrombus Formation (Vascular disorders) | 2 (2)
Vessel Perforation Requiring Treatment (investigational device-related) (Injury, poisoning and procedural complications) | 1 (1)
Vessel Stenosis Requiring Reintervention (Vascular disorders) | 1 (1)
Wound Bleeding or Requiring Debridement (Skin and subcutaneous tissue disorders) | 1 (1)
Wound Infection, New or Worsening (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT03124875/Prot_SAP_001.pdf